CLINICAL TRIAL: NCT05110898
Title: Randomized, Single-Blind, Multicenter, Phase III, Non-Inferiority Clinical Trial to Evaluate the Efficacy and Safety of the Fixed-dose Combination of Olmesartan + Indapamide When Compared to the Isolated Drugs in the Treatment of Hypertension.
Brief Title: Efficacy and Safety Study of the Fixed-dose Combination of Olmesartan + Indapamide When Compared to the Isolated Drugs in the Treatment of Hypertension.
Acronym: OLINDA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainfarma Industria Química e Farmacêutica S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYP 005-21
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-10

CONDITIONS: Hypertension; Hypertension,Essential
Keywords: olmesartan; olmesartan medoxomil; indapamide; hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — olmesartan; Indapamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-dose Olmesartan 20mg/40 mg + Indapamide 1,5 mg (Experimental)
  Interventions: Drug: fixed-dose of olmesartan 20mg/40 mg + indapamide 1,5 mg
- Isolated drugs Olmesartan (20 mg or 40 mg) and Indapamide (1,5 mg) (Active Comparator)
  Interventions: Drug: Isolated drugs Olmesartan (20 mg or 40 mg) and Indapamide (1,5 mg)

INTERVENTIONS:
Drug: fixed-dose of olmesartan 20mg/40 mg + indapamide 1,5 mg — Fixed-dose of Olmesartan 20mg or 40 mg + Indapamide 1,5 mg oral administration, once a day for 12 weeks. Initially, the participant will be treated with Olmesartan 20mg + Indapamide 1,5 mg. If after 6 weeks the diastolic blood pressure is above 90 mmHg, the dose will be changed to fixed dose of Olmesartan 40 mg + Indapamide 1,5 mg.
  Arms: Fixed-dose Olmesartan 20mg/40 mg + Indapamide 1,5 mg
Drug: Isolated drugs Olmesartan (20 mg or 40 mg) and Indapamide (1,5 mg) — Isolated drugs Olmesartan (20 mg or 40 mg) and Indapamide (1,5 mg) oral administration, once a day for 12 weeks. Initially, the participant will be treated with Benicar® (olmesartan) 20mg and Natrilix® (indapamide) 1,5 mg. If after 6 weeks the diastolic blood pressure is above 90 mmHg, the dose of Benicar® (olmesartan) will be changed to 40 mg.
  Arms: Isolated drugs Olmesartan (20 mg or 40 mg) and Indapamide (1,5 mg)

SUMMARY:
Phase III clinical trial, multicenter of non-inferiority, randomized, single-blind evaluation of fixed-dose combination of olmesartan + indapamide compared to the isolated drugs in the treatment of hypertension.

DETAILED DESCRIPTION:
This study is designed for the treatment of essential hypertension. It is performed in participants of both sexes, over 18 years of age, who have essential hypertension with diastolic blood pressure between 90 mmHg and 110 mmHg.

The rationale for studying the fixed dose combination is the possibility to enhance compliance and simplify treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form;
* Participants of both genders aged ≥ 18 years;
* Essential hypertension based on a Diastolic Blood Pressure (DBP) > 90 mmHg and < 110 mmHg;
* Patients with no treatment or on antihypertensive therapy taking up to two anti-hypertensives;
* Possibility of discontinuing previous antihypertensive medication during the washout period.

Exclusion Criteria:

* Essential hypertension based on a Diastolic Blood Pressure (DBP) ≥ 110mmHg and Systolic Blood Pressure (SBP) ≥ 180 mmHg;
* Secondary hypertension;
* Participants with Body Mass Index (BMI) > 35 Kg/m2;
* Non-controlled types 1 and 2 diabetes mellitus (HbA1 > 8,5%);
* Myocardial infarction, coronary surgery or coronary angioplasty with or without stent placement, in the last 6 months;
* Unstable angina;
* Participants with coronary heart disease taking beta-blockers;
* Clinically manifest heart failure;
* History of cardiac arrhythmia;
* Moderate and severe heart valve disease;
* Stroke or transient ischemic attack in the last 6 months;
* Chronic disease of any nature that contraindicates the participant's participation according to the investigator's judgment, in particular renal failure with glomerular filtration rate < 45 ml/min, serum potassium levels ≥ 5,5 mEq/L or ≤ 3,5 mEq/L, hepatopathies, or SGOT, SGPT or bilirubin levels 3 times above the normal upper limit, and blood dyscrasias;
* Known allergies or contraindication to the use of the study medication components;
* Female participants who are pregnant, breastfeeding or who want to become pregnant;
* COVID-19 symptoms;
* Post COVID-19 syndrome with cardiovascular impairment;
* Subjects who have participated in other study within the 12 months prior to screening (unless benefit is justified by the researcher).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of fixed dose association of olmesartan + indapamide compared to the isolated drugs in the treatment of hypertension. | 12 weeks of treatment
  To evaluate the non-inferiority of the fixed dose association of olmesartan + indapamide to the isolated drugs in the change of the diastolic blood pressure from baseline to 12 week endpoint through Ambulatory Blood Pressure Monitoring.

SECONDARY OUTCOMES:
Diastolic Blood Pressure Control | 12 weeks of treatment
  Proportion of participants achieving a diastolic blood pressure below 90 mmHg
Systolic Blood Pressure Control | 12 weeks of treatment
  Proportion of participants achieving a systolic blood pressure below 140 mmHg
Proportion of systolic and diastolic treatment response | 12 weeks of treatment
  Proportion of participants achieving a systolic blood pressure reduction greater than 20 mmHg and a diastolic blood pressure reduction greater than 10 mmHg.
Systolic and diastolic blood pressure variation by ABPM exam | 12 weeks of treatment
  Systolic and diastolic blood pressure variation by ABPM examination from the baseline period compared to the result after 12 weeks of treatment;
Patients responses to the treatment satisfaction questionnaire | 12 weeks of treatment
  Patients responses to a questionnaire regarding if they are satisfied with the treatment.
Tolerability and occurrence of adverse events (AEs) during the study period. | 12 weeks of treatment
  Tolerability and occurrence of adverse events (AEs) during the study period in both study arms.

IPD SHARING:
Plan to Share IPD: No